CLINICAL TRIAL: NCT01629095
Title: Genetic Studies of Non-Alcoholic Fatty Liver Disease
Status: Terminated | Type: Observational
Why Stopped: Slow/insufficient accrual
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120147; 12-HG-0147
Record Dates: First submitted 2012-06-22; First posted 2012-06-27 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Non-Alcoholic Steato-Hepatitis; Liver Cirrhosis; Non-Alcoholic Fatty Liver Disease
Keywords: Liver Transplantation; Genetics
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- NAFLD: Patients who have already undergone liver transplantation for a confirmed diagnosis of NAFLD or cryptogenic cirrhosis are also eligible to participate.
- NASH: Patients with radiologic evidence of fatty liver and/or cirrhosis in which other causes havebeen ruled out are eligible to participate.

SUMMARY:
Background:

- Non-alcoholic fatty liver disease is the most common form of liver disease in the United States. It includes many conditions. Researchers want to study fatty liver disease by looking at people who have liver cirrhosis. They also want to look at people who are or were listed for liver transplants. Genetic studies may provide more information on the causes of these conditions.

Objectives:

- To study possible genetic causes of non-alcoholic fatty liver disease.

Eligibility:

- Individuals of any age who have non-alcoholic fatty liver disease and related conditions.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will provide a blood sample for genetic testing. Liver tissue from a transplant or biopsy may also be studied.
* Participants may also be asked to have an imaging study of the liver. This imaging study may be an x-ray or magnetic resonance imaging.
* No treatment will be provided as part of this research study.

DETAILED DESCRIPTION:
Non-Alcoholic Fatty Liver Disease (NAFLD) is the most common form of liver disease in the United States. It includes a wide spectrum of conditions from benign hepatic steatosis to cirrhosis and liver failure. Non-Alcoholic Steatohepatitis (NASH) is a term that describes specific histological characteristics of liver inflammation and seems to be a determinant step in the progression of NAFLD to cirrhosis and liver failure. The overall purpose of this study is to increase our understanding of the genetic background and pathophysiology of NAFLD through detailed review of physical, radiologic and pathology characteristics, when available. We will perform genetic analysis of known and candidate genes and will assess inheritance through evaluation of unaffected relatives. Most patients will be seen by hepatologists in transplant centers and hepatology clinics across the country. A subset of patients and their families may be seen at the NIH Clinical Center.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Although a liver biopsy is necessary to make the diagnosis of NASH, patients with radiologic evidence of fatty liver and/or cirrhosis in which other causes have been ruled out are eligible to participate.
  2. Patients who have already undergone liver transplantation for a confirmed diagnosis of NAFLD or cryptogenic cirrhosis are also eligible to participate.
  3. Depending on their willingness to participate, subjects may enroll in DNA laboratory-only or clinical-only. However, to conserve resources and meet study objectives, subjects with known pathogenic mutations will be given priority in selection for extensive clinical studies.
  4. Direct blood relatives (typically parents and siblings) of affected individuals with NAFLD and associated conditions are also eligible to participate.

EXCLUSION CRITERIA:

1. Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors) or assent.
2. Pregnant women. Although fatty liver and cirrhosis are sometimes diagnosed during pregnancy, it is unclear if they were present before and just not diagnosed or if they develop as a complication of pregnancy. Additionally energy metabolism changes during pregnancy and lactation which may confound our analysis. If the condition persists after pregnancy and the diagnosis of NAFLD is

   clearly established, patients can be referred to the study.
3. We will review a clinical description from the referring physician about a potential research subject to determine that the subject is appropriate to enter into the study. We reserve the right to exclude cases that are clearly not NAFLD or related to our direct research interests (e.g. fatty liver induced by chronic alcohol use, infectious causes, drug-related, or toxin-related). This almost never happens. However, as some of these environmental factors may contribute to a multifactorial etiology of hepatic changes, we may not exclude all such cases.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Although a liver biopsy is necessary to make the diagnosis of NASH, patients with radiologic evidence of fatty liver and/or cirrhosis in which other causes have been ruled out are eligible to participate. Patients who have already undergone liver transplantation for a confirmed diagnosis of NAFLD orcryptogenic cirrhosis are also eligible to participate.Direct blood relatives (typically parents and siblings) of affected individuals with NAFLD and associated conditions are also eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-04-23 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
To better understand the underlying mechanisms of liver regeneration and the development of NASH. | One point in time
  (a) To determine the role of the Sonic Hedgehog signaling pathway and related genes in the predisposition to liver injury and NASH.(b) To compare gene variants (with known or suspected abnormal functional effects) with the phenotypes observed in patients (i.e. genotype- phenotype correlations) as documented in the study.(c) To verify recurrence risks /inheritance patterns for each of the candidate genes.

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Kruszka, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Transplantation Clinic, Cleveland, Ohio
  - Baylor University Medical Center, Dallas, Texas

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-HG-0147.html